CLINICAL TRIAL: NCT03280771
Title: The Hope Soap Study: a Randomized Controlled Trial of a Hand-washing Intervention Among Children in South Africa
Brief Title: The Hope Soap Study: a Hand-washing Intervention Among Children in South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: Abdul Latif Jameel Poverty Action Lab (Other)
Responsible Party: Principal Investigator, Brendan Maughan-Brown, Senior Research Officer, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1952:BURNSFW
Record Dates: First submitted 2017-09-08; First posted 2017-09-12 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Hand-washing Behavior; Diarrhea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hope Soap group (Experimental): Children in treatment households received a bi-monthly delivery of HOPE SOAP©, a colourful, translucent bar of soap with a toy embedded in its centre
  Interventions: Combination Product: Hope Soap
- Control group (Active Comparator): Children in control households received a colourful, translucent bar or soap with the toy alongside it.
  Interventions: Combination Product: Control group soap

INTERVENTIONS:
Combination Product: Hope Soap — HOPE SOAP© is a colourful, translucent bar of soap with a toy embedded in its centre.
  Arms: Hope Soap group
Combination Product: Control group soap — A colourful, translucent bar or soap with the toy alongside it
  Arms: Control group

SUMMARY:
The Hope Soap Study is a randomised-control pilot study of a hand-washing intervention in which children in treatment households received a bi-monthly delivery of HOPE SOAP©, a colourful, translucent bar of soap with a toy embedded in its centre.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the Family-in-Focus program
* Caregiver provided informed consent
* the age-eligible children were not involved in any other sort of ECD program (e.g. crèche or other day-care)

Exclusion Criteria:

* Enrollment in an ECD program

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 288 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2014-12-15 (Actual); Study Completion 2015-12-15 (Actual)

PRIMARY OUTCOMES:
Direct observation of hand washing prior to eating a snack | 8 weeks
  Hands washed unprompted prior to eating a snack

SECONDARY OUTCOMES:
Questionnaire data on hand washing after using the toilet (scale of 1-10) | 8 weeks
  A score of 1-10 of hand washing after using the toilet
Questionnaire data on hand washing prior to meals (scale of 1-10) | 8 weeks
  A score of 1-10 of hand washing prior to eating meals
Questionnaire data on general soap usage when washing hands (scale of 1-10) | 8 weeks
  A score of 1-10 of soap usage when hands are washed
Questionnaire data on experience of illness (13 items) | 2 weeks
  A score of 1-13 based on self-reported symptoms of illness

REFERENCES:
- [Derived] Burns J, Maughan-Brown B, Mouzinho A. Washing with hope: evidence of improved handwashing among children in South Africa from a pilot study of a novel soap technology. BMC Public Health. 2018 Jun 7;18(1):709. doi: 10.1186/s12889-018-5573-8. PMID 29879942